CLINICAL TRIAL: NCT00415467
Title: Phase IV GliaSite® Radiation Therapy System Registry Protocol for the Treatment of Resectable Malignant Brain Tumors
Brief Title: Treatment of Resectable Malignant Brain Tumors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0942
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Radiation Therapy System; GliaSite RTS
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GliaSite Radiation Therapy System (RTS) (Experimental): Surgical removal of brain tumor followed by GliaSite RTS targeted brachytherapy to the specific brain tumor site
  Interventions: Device: GliaSite Radiation Therapy System

INTERVENTIONS:
Device: GliaSite Radiation Therapy System — Radiation delivery system that provides brachytherapy targeted to a specific site in the brain, to see its effects to the surrounding area where the tumor was located.
  Other Names: GliaSite RTS

SUMMARY:
The goals of this study are to evaluate each of the following items:

1. Time to recurrence in patients receiving brachytherapy with the GliaSite RTS
2. Overall survival (OS) in patients with malignant brain tumors who are undergoing surgical resection and brachytherapy treatment with the GliaSite® Radiation Therapy System (RTS).
3. Incidence of serious adverse events in patients treated with GliaSite RTS

DETAILED DESCRIPTION:
Your doctor has found that you have a brain tumor that needs to be surgically removed. Your doctor has explained the risks and benefits of the surgery. After the brain tumor is surgically removed, some tumor may be left. A treatment that sends additional radiation right to the place around where the tumor was located, may help kill any tumor cells left after the surgery. This treatment is called brachytherapy. Your doctor has explained the risks and benefits of brachytherapy. Researchers in this study would like to evaluate a radiation delivery system, GliaSite RTS, that provides brachytherapy targeted to a specific site in the brain, to see its effects to the surrounding area where the tumor was located.

The GliaSite RTS is a balloon attached to the end of a tube with an access port. The balloon will be put in the space left behind after your tumor is taken out. The end of the tube with its access port will be on the outside of your skull, underneath the skin, at the top of your head. The balloon is filled with radiation therapy solution to provide radiation therapy to any remaining tumor cells next to the space where the tumor was removed.

Before your already scheduled surgery, a series of tests will be performed to find out if you qualify for participation in this study. You will have a complete medical history and your temperature, blood pressure, and pulse will be measured. A standard neurological exam will be performed, in which your mental status, vision, sensory functions, speech, motor skills, and functioning will be evaluated. Women who are able to have children must have a negative urine or blood pregnancy test. A MRI/CT scan will be taken of your head. As part of this MRI/CT, you will get an injection of a contrast solution into your vein. The MRI/CT images will show if there is brain swelling or bleeding. It will also show the edges of the tumor area and will be used to confirm that you should receive radiation therapy with the GliaSite RTS.

If you qualify for the study, you will have a small balloon (GliaSite) placed in the space where the tumor was removed during your surgery. The balloon will be filled with an x-ray dye and normal saline (sterile water with salt) to make sure that the balloon properly fills the space where the tumor was removed. Your surgeon will then stitch your head closed. It is possible that your surgeon may decide not to place the GliaSite device in the space where the tumor was. If your surgeon chooses not to place the GliaSite device, you will be offered alternative treatments, once you recover from surgery.

The balloon will be filled with an x-ray dye solution once it has been placed in the surgical cavity and will be kept filled until it is replaced by the radioactive solution. You will then have an MRI/CT of the head. Following this MRI/CT exam, you will get an injection of a contrast solution into your vein. You will then have a second MRI/CT exam of the head, which will show this contrast solution. The MRI/CT images will show if there is brain swelling or bleeding. It will also show the edges of the tumor area and where the balloon is located. These images will be used to confirm that you should receive radiation therapy with the GliaSite RTS device. You may also have x-ray films of the brain to confirm balloon placement. You may be able to leave the hospital after surgery.

You may be readmitted to the hospital for radiation therapy about one to two weeks after surgery. Twenty-four hours before starting radiation therapy, you will begin taking a medication and continue taking it for 24 hours after your radiation therapy is finished. This medication, an iodine-potassium iodide solution, keeps your thyroid gland from gathering too much radiation in the event that the balloon leaks.

Before the radiation therapy is begun, x-ray films of the brain may be taken to show the location of the balloon and verify the balloon is still properly placed. Once the placement of the balloon is confirmed, the x-ray dye and saline are removed from the catheter. The balloon will then be filled with radiation therapy solution and normal saline.

You may be able to go home once the material has been put into the balloon. If this is done, special instructions will be given to you that you must follow if you are sent home. You must then return to the hospital at the appropriate time for removal of the radioactive material. Otherwise, you will be in the hospital the entire time you are getting radiation therapy.

When the radiation therapy is completed after about 3 to 7 days, the radiation therapy solution will be removed from the balloon. The GliaSite device will be rinsed with normal saline. This rinsing helps lessen any radioactivity remaining in the device. After completion of brachytherapy, the balloon will be completely emptied and the GliaSite device will be surgically removed. When your doctor feels that you are ready, you will be discharged from the hospital.

Following the completion of brachytherapy, you may receive other forms of radiation therapy as prescribed by your physician. This is usually done as an outpatient.

You will be asked to follow up with your doctor at certain time points after you receive the brachytherapy treatment. The time points are 1 month and 3 months after brachytherapy and then every 3 months after that (for example, 1, 3, 6, 9, 12, 15, 18, 21 and 24 months).

During these follow up visits, you will be asked to complete a mini-mental status examination referred to as a MMSE. You will be asked to complete a quality of life questionnaire. Your physician may take an MRI or CT image of your brain if he/she thinks it is necessary.If you have undergone a second operation for your brain cancer, you will be asked about this surgery. You will be asked about any steroid medication you are taking and if the dose has changed since your last visit. Your doctor will also ask you about any other cancer medications or treatments you have received since your last visit.You and your doctor may discuss any serious events that have happened to you since your last visit.

This is an investigational study. The device is FDA approved. About 300 patients will take part in this multicenter study. Up to 20 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically proven malignant brain tumor
2. Patient must be a candidate for surgical resection of the tumor mass.
3. Patient must not be pregnant or breast-feeding. All patients with the potential for pregnancy should be counseled and requested to follow acceptable birth control methods to avoid conception.
4. Patient must sign informed consent form

Exclusion Criteria:

1. Serious concurrent infection or medical illness which could jeopardize the ability of the patient to receive the GliaSite catheter with reasonable safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to Recurrence of Brain Tumor (anywhere in brain) | From brachytherapy to assessments at 1 and 3 months after brachytherapy then every 3 months after that or until documented brain tumor recurrence.
  Time to recurrence of brain tumor determined for each patient from the time at the end date of brachytherapy with the GliaSite RTS until the date of documented brain tumor recurrence.

SECONDARY OUTCOMES:
Overall Patient Survival | Time from completion of the GliaSite procedure to death by any cause (time in months).
  Overall survival determined as time from end date of brachytherapy with the GliaSite RTS until the date of death, including occurrences of death due to CNS causes and by deaths due to non-CNS causes. In the time to event analyses, if the event is not reached, participant censored at last date known to be without the event of interest (recurrence-free or alive). Median time-to-event determined by Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Mahajan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org